CLINICAL TRIAL: NCT02351934
Title: A Prospective, Randomized Study Evaluating the Efficacy and Safety of Early Diuresis Following Colorectal Surgery
Brief Title: Early Diuresis Following Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ilya M. Danelich, Pharm.D., R.Ph., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-008292; UL1TR000135 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-01-30 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Disorders
Keywords: colorectal surgery; volume status
MeSH Terms: interventions — Furosemide; Celecoxib; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Furosemide + Enhanced Recovery after Surgery (ERAS) (Experimental): Furosemide 10 mg IV on post-operative day #1 and/or 2, plus ERAS, as described in other arm.
  Interventions: Drug: Furosemide; Drug: Celecoxib; Drug: Gabapentin
- Enhanced Recovery after Surgery (ERAS) (Active Comparator): ERAS included administration of celecoxib and gabapentin in the pre-operative setting, single-injection intrathecal analgesic administration immediately prior to induction of general anesthesia, post-operative administration of scheduled acetaminophen and nonsteroidal anti-inflammatory drug (NSAID) or tramadol, and discontinuation of IV fluids by 0800 on postoperative day (POD) 1. Intraoperative fluid administration was dependent on the individual anesthesia provider with no unified commitment to either zero balance or goal-directed fluid therapy. Fluid status was determined based on patient weight. Patients were weighed preoperatively and daily post-operatively using either a bed scale or a unit-based scale.
  Interventions: Drug: Celecoxib; Drug: Gabapentin

INTERVENTIONS:
Drug: Furosemide
  Other Names: Lasix
  Arms: Furosemide + Enhanced Recovery after Surgery (ERAS)
Drug: Celecoxib — Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) used to treat pain or inflammation.
  Other Names: Celebrex
Drug: Gabapentin — Gabapentin is a oral drug used to treat seizures, postherpetic neuralgia, and restless legs syndrome.
  Other Names: Neurontin

SUMMARY:
The purpose of this study is to find out if giving a medicine called furosemide, which is a diuretic or water pill, after colon surgery will safely shorten the patient's length of hospital stay.

DETAILED DESCRIPTION:
This study will assess if administration of a loop diuretic, specifically furosemide, to achieve euvolemia can safely reduce length of stay following colorectal surgery.

ELIGIBILITY:
Inclusion Criteria

* All elective colorectal surgeries (CRS) utilizing the enhanced recovery pathway (ERP)
* The surgery involves resection

Exclusion Criteria

Exclusion Criteria for Randomization:

* Surgeries involving intraoperative radiation
* Ileostomy closures, when performed as the only surgical intervention
* Surgeries involving multiple disciplines (e.g., colorectal plus general surgery, colorectal plus gynecology surgery) except for colorectal surgeries plus ureteral stent placements.
* Chronic loop diuretic therapy (i.e., bumetanide, torsemide, furosemide, ethacrynic acid) including as needed administration of such therapy
* Patients receiving dialysis
* Creatinine clearance, calculated by the Cockcroft-Gault equation, less than 30 mL/min.
* Inpatient prior to surgery
* Allergy to furosemide
* Allergy to sulfa drugs if the allergy involves anaphylactic reaction
* Lack of serum creatinine concentration within 3 months preceding the surgery AND diagnosis of chronic kidney disease

Exclusion Criteria for Intervention (applies to both the intervention and control arm):

* Patient's weight on postoperative day (POD) #1 and POD #2 is less than preoperative weight.
* Blood pressure criteria: systolic blood pressure criteria less than 90 mmHg or greater than 30 mmHg below baseline on POD #1 and/or POD #2 immediately prior to administration of study drug.
* Complications within 48 hours of surgery
* Abscess (infected fluid collection, treated with CT drainage)
* Leak (defined by CT drainage or reoperation)
* Wound infection (treated with either antibiotics and/or open packing)
* Bowel obstruction (treated with reoperation)
* Reoperation
* Hemorrhage
* Weight change since admission on POD #1: > 5 kg
* Acute kidney injury on POD #1 and POD#2 defined as serum creatinine (SCr) increase ≥ 0.3 mg/dL or increase to ≥ 150% to 200% (1.5- to 2-fold) from baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Danelich, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota between February 2015 and April 2016.
Period: Allocation
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Started | 62 | 61
Received Allocation | 56 | 61
Completed | 56 | 61
Not Completed | 6 | 0
Not completed — POD weight<pre-op weight | 3 | 0
Not completed — Hypotension preventing administration | 2 | 0
Not completed — Acute Kidney Injury on Post Op Day 1 | 1 | 0
Period: Follow-Up
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Started | 56 | 61
Completed | 44 | 51
Not Completed | 12 | 10
Not completed — POD weight<pre-op weight | 3 | 0
Not completed — Acute Kidney Injury | 1 | 0
Not completed — Early dismissal | 3 | 0
Not completed — Hypotension | 3 | 0
Not completed — No documentation | 2 | 0
Not completed — 1 ERAS Component Noncompliant | 0 | 6
Not completed — 2 ERAS Components Noncompliant | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS) | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [42 to 68] | 61 [45 to 68] | 59 [42 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 40 | 33 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 61 | 123

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Participants will be followed for the duration of hospital stay, an expected average of 2-7 days.
Time Frame: Up to 7 days
Population: Intent to treat analysis
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
hours | 99.6 [73.1 to 150.6] | 80.6 [73.6 to 124.0]
Statistical Analysis 1: Comparison: Furosemide + Enhanced Recovery After Surgery (ERAS) vs Enhanced Recovery After Surgery (ERAS); Significance level of 0.05 was used; Test type: Superiority; p = 0.564, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants Readmitted to Mayo Clinic Within 30-days
Time Frame: Within 30 days of release from hospital
Population: Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
Participants | 13 | 10
Statistical Analysis 1: Comparison: Furosemide + Enhanced Recovery After Surgery (ERAS) vs Enhanced Recovery After Surgery (ERAS); Significance level of 0.05 was used; Test type: Superiority; p = 0.675, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants Requiring Nasogastric Tube Placement
Time Frame: Up to 7 days
Population: Intention to Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
Participants | 6 | 1
Statistical Analysis 1: Comparison: Furosemide + Enhanced Recovery After Surgery (ERAS) vs Enhanced Recovery After Surgery (ERAS); Significance level of 0.05 was used; Test type: Superiority; p = 0.125, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time to Stool Output
Time Frame: Up to 4 days
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
hours | 48.8 [27.8 to 82.2] | 45.4 [22.7 to 68.8]

5. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Acute kidney injury (AKI) refers to an abrupt decrease in kidney function, resulting in the retention of urea and other nitrogenous waste products and in the dysregulation of extracellular volume and electrolytes. The term AKI has largely replaced acute renal failure (ARF), reflecting the recognition that smaller decrements in kidney function that do not result in overt organ failure are of substantial clinical relevance and are associated with increased morbidity and mortality. The AKI experienced by these patients was not considered an adverse event.
Time Frame: Up to 7 days
Population: Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
Participants | 2 | 2
Statistical Analysis 1: Comparison: Furosemide + Enhanced Recovery After Surgery (ERAS) vs Enhanced Recovery After Surgery (ERAS); Significance level of 0.05 was used; Test type: Superiority; p = 0.595, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Hypokalemia
Description: Hypokalemia is generally defined as a serum potassium level of less than 3.5 mmol/L.
Time Frame: Up to 7 days
Population: Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
Number analyzed (Participants) | 62 | 61
Participants | 2 | 3
Statistical Analysis 1: Comparison: Furosemide + Enhanced Recovery After Surgery (ERAS) vs Enhanced Recovery After Surgery (ERAS); Significance level of 0.05 was used; Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Furosemide + Enhanced Recovery After Surgery (ERAS) | Enhanced Recovery After Surgery (ERAS)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 8/62 | 3/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide + Enhanced Recovery After Surgery (ERAS) (N=62) | Enhanced Recovery After Surgery (ERAS) (N=61)
Decreased Potassium (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Increased Serum Creatinine (Renal and urinary disorders) | 2 (2) | 0 (0) — If your kidneys aren't functioning properly, an increased level of creatinine may accumulate in your blood.
Decreased blood pressure (Cardiac disorders) | 3 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Urine leak (Renal and urinary disorders) | 0 (0) | 1 (1)
Increased heart rate (Cardiac disorders) | 1 (1) | 0 (0)
Increased temperature (General disorders) | 1 (1) | 0 (0)
Hematoma/Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes